CLINICAL TRIAL: NCT06114472
Title: The Impact of Preoperative Aromatherapy Upon Time to First Analgesia Request and Consumption After Cesarean Section; Randomized Clinical Trial
Brief Title: The Impact of Preoperative Aromatherapy Upon Time to First Analgesia Request After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB8888888888
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A aromatherapy (Active Comparator): three drops of aromatherapy blend containing Lavender essence 10% were poured on cotton in cast containers, and the patient was asked to inhale it for 5 minutes from a distance of 10 cm
  Interventions: Drug: aromatherapy blend containing Lavender
- Group B Control (No Intervention): No intervention

INTERVENTIONS:
Drug: aromatherapy blend containing Lavender — hree drops of aromatherapy blend containing Lavender essence 10% were poured on cotton in cast containers, and the patient was asked to inhale it for 5 minutes from a distance of 10 cm
  Arms: Group A aromatherapy

SUMMARY:
one of the main aims of anesthesia is to reduce postoperative pain. However, many drugs that are used for this purpose, especially opioids, have side effects such as respiratory distress, nausea, itching, and gastrointestinal bleeding

. Recent studies have indicated interest in using complementary therapies such as heat and cold therapy, hypnotism.

DETAILED DESCRIPTION:
Pain is amongst the most common problems after surgery

(1). Pain is an unpleasant sensory and emotional experience, which is associated with the real or probably damage of tissue. Unrelieved postoperative pain in addition to creating fears in the surgical patients, it makes adverse psychological impact on them

* The uncontrolled postoperative pain will make a lot of acute and chronic effects, including systemic mediators, hypercoagulability, postoperative immunosuppression, and delayed wound healing
* So, one of the main aims of anesthesia is to reduce postoperative pain. However, many drugs that are used for this purpose, especially opioids, have side effects such as respiratory distress, nausea, itching, and gastrointestinal bleeding. Recent studies have indicated interest in using complementary therapies such as heat and cold therapy, hypnotism.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 40 years
* Body mass index (BMI) of 18-35 kg/m2
* Patients with the American Society of Anesthesiologists (ASA) physical status I/II,
* Patients scheduled for elective cesarean section.

Exclusion Criteria:

* Patient refusal

  * Allergy to local anaesthetics
  * Anosmia
  * Coagulopathy,
  * Chronic pain syndromes
  * Prolonged opioid medication
  * Patients who received any analgesic 24 h before surgery.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
time to first analgesia request | 24 hours
  time to first analgesia request in minutes

SECONDARY OUTCOMES:
Total daily consumption of analgesia | 24 hours
  intravenous keteloac total consumption in the 1st 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McQuay H, Derry S, Wiffen P, Moore A, Eccleston C. Postoperative pain management: number-needed-to-treat approach versus procedure-specific pain management approach. Pain. 2013 Jan;154(1):180. doi: 10.1016/j.pain.2012.10.007. Epub 2012 Oct 22. No abstract available. PMID 23200259
- [Background] Gupta A, Kaur K, Sharma S, Goyal S, Arora S, Murthy RS. Clinical aspects of acute post-operative pain management & its assessment. J Adv Pharm Technol Res. 2010 Apr;1(2):97-108. PMID 22247838
- [Background] Sheikhan F, Jahdi F, Khoei EM, Shamsalizadeh N, Sheikhan M, Haghani H. Episiotomy pain relief: Use of Lavender oil essence in primiparous Iranian women. Complement Ther Clin Pract. 2012 Feb;18(1):66-70. doi: 10.1016/j.ctcp.2011.02.003. Epub 2011 Mar 16. PMID 22196577